CLINICAL TRIAL: NCT06457828
Title: Effect of Apical Patency and Local Corticosteroid on Pain and Neuropeptides Release in Patients With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mustafa M. Sultan, Teaching assistant, Suez Canal University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 291/2020
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain; Symptomatic Irreversible Pulpitis
Keywords: Pulpitis; Postoperative Pain; VAS
MeSH Terms: conditions — Pain, Postoperative; Pulpitis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No apical patency (Sham Comparator)
  Interventions: Procedure: Non-corticosteroid injection; Drug: Corticosteroid injection
- Apical patency (Active Comparator)
  Interventions: Procedure: Non-corticosteroid injection; Drug: Corticosteroid injection

INTERVENTIONS:
Procedure: Non-corticosteroid injection — no infiltration injection of 0.7 ml of dexamethasone lateral to the involved tooth after anesthesia administration.
Drug: Corticosteroid injection — infiltration injection of 0.7 ml of dexamethasone lateral to the involved tooth after anesthesia administration.

SUMMARY:
The goal of this randomized clinical trial is to learn the effect of using local corticosteroids and maintaining apical patency in reducing post-preparation pain in patients with acute irreversible pulpitis in molar teeth. The main question it aims to answer is:

• How effective are using local corticosteroids and maintaining apical patency in reducing post-preparation pain in patients with acute irreversible pulpitis? Participants will be asked to fill a visual analogue scale to record their pain, after receiving a root canal treatment while using local corticosteroids or not as well as maintaining apical patency or not.

Researchers will compare the use of corticosteroids and maintaining apical patency in reducing post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic acute irreversible pulpitis in molar teeth.
* Normal periapical condition including periapical radiography with minimal widening of periodontal ligament.
* Normal probing depth.
* No medical condition.
* No contraindication for administration of corticosteroids and local anesthesia.

Exclusion Criteria:

* Facial or oral paresthesia.
* Pregnancy & breastfeeding.
* Unrestorable tooth.
* Marginal periodontal disease.
* Presence of a crown on the tooth involved.
* Over instrumentation during root canal treatment.
* Long-term use of corticosteroids.
* False-positive cases of sensibility test with necrosis discovered after gaining access to the tooth.
* Cases requiring intrapulpal injection to promote anesthesia.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 6, 12, 24, 48, 72 hour and 7 days postoperative intervals
  Patients were instructed to record their pain level using the Visual Analog Scale
Inflammatory markers | before treatment, after 3 days and after 7 days
  Gingival crevicular fluid samples were collected by periopaper for testing the level of IL-1β and IL-10

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt